CLINICAL TRIAL: NCT07368816
Title: Oxygen-enriched Oil-based Dressing: a New Option for Tunneling Post-surgical Diabetic Foot Ulcers
Brief Title: OEOd-Based Wound Dressing in Post-Surgical Diabetic Foot Ulcers
Acronym: OEOd-DFU-pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Alessia Scatena, Diabetologist, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OEOd-AR-38235; OEOd-AR-38235 (Other: Ethics Committee of the Tuscany Region, South-East Area)
Record Dates: First submitted 2026-01-08; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot; Postoperative Wound Healing
Keywords: diabetic foot; wound healing; postoperative wound; pilot study; oxygen-enriched oil-based dressing
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in parallel to one of two study groups: an intervention group receiving an OEOd-based wound dressing and a control group receiving standard wound care. Each participant was allocated to a single treatment group for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OEOd-Based Wound Dressing (Experimental): Participants assigned to this arm received a topical OEOd-based wound dressing applied to post-surgical diabetic foot ulcers according to routine clinical practice, in addition to standard multidisciplinary diabetic foot care.
  Interventions: Device: OEOd-based wound dressing
- standard wound care (Active Comparator): Participants assigned to this arm received standard wound care for post-surgical diabetic foot ulcers according to institutional clinical practice.
  Interventions: Other: Standard of Care (Investigator Choice)

INTERVENTIONS:
Device: OEOd-based wound dressing — Topical application of an OEOd-based wound dressing to post-surgical diabetic foot ulcers according to routine clinical practice, in addition to standard multidisciplinary diabetic foot care.
  Arms: OEOd-Based Wound Dressing
Other: Standard of Care (Investigator Choice) — Conventional wound management for post-surgical diabetic foot ulcers according to institutional standard clinical practice.
  Arms: standard wound care

SUMMARY:
This study is a prospective randomized controlled pilot study evaluating the efficacy and safety of an OEOd-based wound dressing compared with standard wound care in patients with post-surgical diabetic foot ulcers. Participants were randomly assigned at enrollment to receive either the OEOd-based dressing or standard therapy. The primary outcome was complete ulcer healing at 16 weeks. Secondary outcomes included new infections, need for additional surgical debridement, re-hospitalization, and time to healing. The study was designed to provide preliminary estimates of treatment effect and feasibility to inform future larger randomized trials.

DETAILED DESCRIPTION:
This study was designed as a prospective randomized controlled pilot study to evaluate the efficacy and safety of an OEOd-based wound dressing compared with standard wound care in patients with post-surgical diabetic foot ulcers. Adult patients with diabetes mellitus presenting with a post-surgical foot ulcer were prospectively enrolled and randomly assigned at the time of enrollment to receive either the OEOd-based wound dressing or standard therapy, according to a simple random allocation procedure.

All patients received standard multidisciplinary diabetic foot care, including surgical management when indicated, infection control, off-loading, and metabolic optimization. The investigational intervention consisted of a topical OEOd-based wound dressing applied according to routine clinical practice.

The primary endpoint of the study was complete ulcer healing at 16 weeks, defined as full epithelialization of the target lesion without drainage. Secondary endpoints included the occurrence of new infections, the need for additional surgical debridement, re-hospitalization during follow-up, and time to healing, which was evaluated as an exploratory outcome.

Given the pilot nature of the study, no formal a priori sample size calculation was performed. The trial was intended to provide preliminary estimates of treatment effect and feasibility to inform the design of future larger randomized controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with diabetes mellitus
* Presence of a post-surgical diabetic foot ulcer
* Eligibility for topical wound treatment
* Ability to provide written informed consent

Exclusion Criteria:

* Active malignancy
* Severe systemic infection or sepsis
* Known hypersensitivity to components of the wound dressing
* Inability to comply with study procedures or follow-up
* Participation in another interventional clinical study during the same period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Complete ulcer healing | 16 weeks
  number of ulcers completely healed at 16 weeks

SECONDARY OUTCOMES:
new infections | 16 weeks
  number of patients with new clinically diagnosed wound infections during follow-up.
Additional surgical debridement | 16 weeks
  number of patients needing additional surgical debridement of the target ulcer during follow-up.
re-hospitalization | 16 weeks
  number of Hospital admission related to the target ulcer during the follow-up period.
time to healing | 16 weeks
  Time from enrollment to complete ulcer healing, evaluated as an exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Scatena, MD, Principal Investigator — Diabetology and Metabolism Unit, San Donato Hospital Arezzo, Local Health Authority South-East Tuscany, iTaly
Locations (1):
- Diabetology and Metabolism Unit, San Donato Hospital Arezzo, Local Health Authority South-East Tuscany, iTaly, Arezzo, AR, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the pilot nature of the study and to protect patient confidentiality.

REFERENCES:
- [Result] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- See also: key reference on the clinical management of diabetic foot ulcers — https://pubmed.ncbi.nlm.nih.gov/28614674/